CLINICAL TRIAL: NCT06614647
Title: RESPONSE: Colorectal Cancer Survivors' Follow-up Care - Now Digital and Need-based: A National Interventional Effectiveness Trial for Stage I and II Patients
Brief Title: RESPONSE: Colorectal Cancer Survivors' Follow-up Care - Now Digital and Need-based
Acronym: RESPONSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); University of Southern Denmark (Other); Randers Regional Hospital (Other); Viborg Regional Hospital (Other); Gødstrup Hospital (Other); Odense University Hospital (Other); Herlev Hospital (Other); Bispebjerg Hospital (Other); Sygehus Lillebaelt (Other); Svendborg Hospital (Other)
Responsible Party: Principal Investigator, Claus Lindbjerg Andersen, Professor, Group Leader, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RESPONSE
Record Dates: First submitted 2024-07-09; First posted 2024-09-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Quality of Life; Survivorship
Keywords: Circulating Tumor DNA; Organ-specific late effects; Biopsychosocial Late effects
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The region of residency determines the allocation to the intervention group or standard-of-care group. Patients in the intervention group will be stage I-II colorectal cancer survivors residing in Central Denmark Region and North Denmark Region. Both regions have fully implemented 'organ-specific late-effects clinics' offering a standardized patient-centered, interdisciplinary, multiorgan approach and have implemented the digital platform that supports the smartphone care guide. Patients in the standard group will be the corresponding patients residing in the remaining Danish Regions, in which similar standardized late effects clinics and the digital care-guide framework are not yet implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): Patients with curatively resected stage I or low risk stage II colorectal cancer, residing in Central or North region, Denmark.
  Interventions: Diagnostic Test: Recurrence monitoring with circulating tumor DNA (ctDNA) as a high risk biomarker; Behavioral: Monitoring for late adverse effects with electronic patient reported outcome measures (ePROMs); Behavioral: Systematic treatment of organ-specific late effects and/or biopsychosocial late effects; Behavioral: Digital care-guide for long-term follow-up after cancer treatment
- Standard-of-care group (SG) (No Intervention): Patients with curatively resected stage I or low risk stage II colorectal cancer, residing in South or Capital region, Denmark.

INTERVENTIONS:
Diagnostic Test: Recurrence monitoring with circulating tumor DNA (ctDNA) as a high risk biomarker — IG patients will receive the following intervention at 3, 12, 24, and 36 months post-surgery:
  1) Recurrence risk stratification by ctDNA analysis of blood samples:
  a) Only if ctDNA becomes positive, will imaging be performed. b) If ctDNA is positive, but recurrent disease is not detected by imaging or clinical and endoscopic evaluation, the patient will be referred back to intensified ctDNA measurements repeated every 4 months until either ctDNA becomes negative or recurrence is confirmed by subsequent imaging.
  Arms: Intervention group (IG)
Behavioral: Monitoring for late adverse effects with electronic patient reported outcome measures (ePROMs) — 2) Collection and analyses of ePROMs to identify whether patients suffer from organ-specific late effects or biopsychosocial late effects and monitor of health related quality of life and the impact of late adverse effects hereon.
  Arms: Intervention group (IG)
Behavioral: Systematic treatment of organ-specific late effects and/or biopsychosocial late effects — 3) When needed, standardized treatment for organ-specific late effects according to newly published national guidelines at specialized centers. Further, online cognitive behavioral therapy is offered to patients suffering from severe biopsychosocial late effects.
  Arms: Intervention group (IG)
Behavioral: Digital care-guide for long-term follow-up after cancer treatment — Use of a digital care-guide from study inclusion to guide the patient trough the follow-up program, in the form of a personalized smart phone app.
  Arms: Intervention group (IG)

SUMMARY:
Over the last decades, the 3-year recurrence rates for patients with stage I and II colorectal cancer have decreased to just 5% and 12%. The follow-up program offered to stage I and low-risk stage II patients has not changed accordingly and is still focused solely on recurrence detection. Moreover, it is a one-size-fits-all program, i.e. most of the follow-up resources are spent on non-recurrence patients who do not benefit.

Up to 50% of cancer survivors suffer from reduced quality of life related to fear of cancer recurrence, treatment-related psychological distress, and/or severe late adverse effects of a biopsychosocial and/or organ-specific origin. Today many of these symptoms can be treated effectively. However, no systematic program aimed at monitoring and addressing the symptoms has been implemented yet.

The current project is testing a newly developed, digitally managed, patient-centered follow-up program that focuses on individual patient needs, including fear of cancer recurrence, psychological well-being, management of late adverse effects, and recurrence surveillance. This new program will be compared to the current standard of care in a national network of 11 colorectal cancer surgical centers in four of five Danish regions.

Patients in the intervention group will receive the following:

1. Risk-stratified circulating tumor DNA (ctDNA) guided recurrence surveillance.
2. Late adverse effects monitoring with electronic patient-reported outcome measures, which are validated questionnaires that can identify and qualify late adverse effects.
3. Systematic treatment for organ-specific and/or biopsychosocial late adverse effects.
4. A digital care guide, to support the patient trajectory through the follow-up program, as a smartphone app.

Patients in the standard group will receive standard-of-care follow-up.

The primary study endpoint will be the difference in health-related quality of life between the intervention and standard group. Secondary outcomes include e.g., comparison of health-related costs, differences in fear of cancer recurrence, recurrence-free survival, and patient satisfaction.

The investigators expect the new follow-up program to be better than the standard-of-care program in terms of the primary endpoint - quality of life - without compromising recurrence detection, and without increasing costs.

DETAILED DESCRIPTION:
Background:

Colorectal cancer (CRC) screening was implemented in Denmark in 2014 and has effectively shifted the CRC stage at the time of diagnosis from late stage (III and IV) to earlier stages (I and II)[1]. Consequently, more patients are offered curative intended treatment, which increases the number of survivors in postoperative follow-up care: In 2020, 65% of Danish patients with CRC, potentially eligible for follow-up care, had stage I-II disease[1].

The current follow-up for CRC survivors is recurrence-focused, with computed tomography (CT) imaging at 12 and 36 months[2] as early recurrence detection is critical to increase the possibility of curative treatment: The 5-year survival rate for patients treated for recurrence with curative intent is ~40% compared to <10% for patients managed with palliative or best supportive care[3-6]. However, the risk of recurrence strongly depends on the CRC stage: The 3-year cumulative recurrence rate is only 4.5%-7.9% for stage I and 10%-16% for stage II[7-9]. Consequently, the resources allocated to CRC follow-up in Denmark are primarily dissipated on patients who will never experience a recurrence. Hence, the challenge remains to distinguish between high- and low-risk patients, i.e., tailor the follow-up program to the personal risk of recurrence instead of "one-size-fits-all".

A promising and novel surveillance method for CRC recurrence is to screen longitudinally collected blood samples for the presence of circulating tumor DNA (ctDNA). Serial ctDNA analyses detect recurrence with high sensitivity (88%) and specificity (97%) independent of the stage (hazard ratio (HR)=40.7; 95% confidence interval (CI): 11.6-143) and with a median lead-time of 7-10 months compared to current standard-of-care follow-up[10-13]. Thus, serial ctDNA analyses have the potential to efficiently identify the 4.5%-16% of stage I-II patients, who should be offered CT imaging, whereas the remaining 84-95% of patients are spared unnecessary CT imaging.

CRC survivors with a low risk of recurrence may perceive other challenges than CRC recurrence as equally or more important in everyday life. Such challenges may include the psychological distress related to the CRC diagnosis, exaggerated fear of cancer recurrence (FCR) regardless of the actual risk of recurrence, and the presence of treatment-related organ-specific late effects, which may negatively impact their quality of life (QoL). Independently of stage, 13% of patients with CRC report persistently low QoL and/or high levels of psychological distress, e.g., impaired emotional well-being and/or high FCR[14].

Approximately half of CRC survivors suffer from organ-specific late effects, e.g., bowel, urinary, or sexual dysfunction[15-18]. In a recent study, 20% of colon cancer patients and 30% of rectal cancer patients expressed a wish for help managing their organ-specific late effects[19]. Besides organ-specific late effects, many CRC survivors experience one or more persistent general symptoms and late effects after their cancer treatment including psychological distress, depression, anxiety, insomnia, fatigue, pain, and impaired cognitive function. While the management of these so-called biopsychosocial late effects has received only little attention until recently, a growing body of evidence suggests that these issues can be treated effectively with cognitive behavioral approaches[20-24]. However, none of these challenges are addressed by today's recommended follow-up care program.

To improve the management of follow-up care, recent studies have demonstrated the benefit of high patient satisfaction with electronic Patient-Reported Outcome Measures (ePROMs)[25]. Furthermore, it has been shown that 80% of Danish patients with CRC respond to ePROMs and that those with organ-specific late effects and/or biopsychosocial late effects can effectively be identified using ePROMs[19]. Hence, ePROMs have the potential to help clinicians stratify CRC survivors to postoperative surveillance or interventions for treating both organ-specific late effects and biopsychosocial late effects.

New technology further facilitates the management of follow-up care: the use of digital care-guides has become increasingly popular in the Danish Health care system. One example is a framework based on a smartphone app that enables implementation of a comprehensive digital care guide in the follow-up program for CRC (Emento)[26]. This app can help maintain patient autonomy, acting as both a reference work and a timed tool to inform, educate, and guide the patient through the follow-up program.

RESPONSE proposes to use each of the elements described above in a new, individualized follow-up program for CRC. All elements have already been tested and have shown their great potential in separate efficacy trials[11-13,19,23,25]. However, the impact of combining all four elements in a single follow-up program has never previously been investigated.

Aim:

The overall aim of this study was to investigate whether the combination of the above elements in recurrence surveillance, could improve health-related QoL (HRQoL), without compromising overall survival (OS) and recurrence-free survival (RFS) or increasing costs. Thus, our study objective was to design a surveillance program fulfilling these criteria. Further, the objective was to conduct a trial where this program could be compared to standard-of-care recurrence surveillance.

The new follow-up program includes: 1) serial ctDNA monitoring to identify individuals with high risk of recurrence, 2) serial ePROMs monitoring to identify 'organ-specific late effects' and 'biopsychosocial late effects', 3) planned and systematic management/intervention of recurrence and late effects, and 4) personalized self-managed follow-up by a digital care guide as a smartphone application.

Study design:

This new program will be compared to the standard-of-care imaging-based recurrence surveillance in a Danish multicenter, interventional effectiveness trial, including 392 patients from 11 surgical centers. The patients will be divided into two arms: the intervention group (IG) and the standard-of-care group (SG).

IG patients (n=196) will receive all the following at 3-,12-,24-, and 36-months post-surgery:

1. Recurrence risk stratification by plasma ctDNA.

   1. If ctDNA becomes positive, CT imaging of the thorax and abdomen will be performed. This enables the CT imaging resources to be directed at the high-risk individuals (=ctDNA positive) only.
   2. The results of the CT imaging are discussed at the usual MDT at the responsible surgical department, where pathologists, oncologists, CRC surgeons, and radiologists are present. The MDT decides whether further diagnostic initiatives should be taken, e.g., endoscopy or further imaging.
   3. If recurrent disease is detected, the patient is treated according to the national Danish guidelines, and the outcome is registered in the RESPONSE trial.
   4. If a recurrence is NOT detected by imaging or subsequent clinical examinations, the patient returns to the RESPONSE trial with increased ctDNA testing frequency every four months.
   5. If longitudinal ctDNA tests become negative, the patient returns to the default ctDNA test frequency.
   6. If longitudinal ctDNA tests are repeatedly positive, CT imaging will be prompted and discussed at MDT until a site of recurrence can be confirmed.
2. Personalized self-managed follow-up care, using a digital platform with longitudinal collection of ePROMs to identify

   1. whether patients suffer from organ-specific late effects and/or biopsychosocial late effects
   2. whether this impacts patients' overall HRQoL.
3. Intervention for organ-specific late effects and/or biopsychosocial late effects if needed.

SG patients (n=196) will receive standard follow-up with CT imaging at 12- and 36-months post-surgery, at the surgical departments according to Danish national guidelines. Any local variation/addition to the standard follow-up program will be allowed.

All SG patients will have longitudinal blood samples collected at the same time points as IG patients but only analyzed after the end of the trial, to enable comparison of ctDNA vs. CT imaging as a recurrence predictor. Furthermore, SG patients will receive similar ePROMs as IG patients to collect information at the same time points. However, these will only be analyzed after the end of the trial.

Outcomes and power calculation:

The primary study outcome will be the difference in HRQoL between groups. This will be calculated as the difference in EORTC-QLQ-C30 (global health/QoL domain) between IG and SG at 36 months.

A mean global score of 61 points in the SG is assumed. A score difference of 7 or more between groups will be considered as the minimal clinical important difference (MID). Thus, 170 patients are required in each group to detect an increase of 7 for a mean global score of 68 in the IG with 80% power and 5% significance level. Expecting a drop-out rate of 10%, 189 patients need to be included in each group.

For the secondary objective, OS and RFS, the difference in cumulative RFS and OS between groups will be calculated at 3 and 5 years. Expectantly the cumulative RFS will be 93% in the SG and 92% in the IG. With 196 patients in each group, a decrease in RFS of 9% in IG can be shown with 80% power at a 5% significance level. Thus, the number of included patients is increased to 196 in each group. Non-inferiority will be declared if the difference in RFS is within this limit. The mean OS in the groups is expectantly 77,5%. With 196 patients in each group, an increase of 10% in OS for the IG can be shown with 70% power at a 5% significance level.

Data analyses and statistics:

All data will be presented using descriptive statistics. The ePROM scores will be calculated according to the scoring guidelines for each of the questionnaires. Missing PRO data in form of missing items within an ePROM assessment will be imputed according to the questionnaire's scoring guideline.

The incremental cost-effectiveness ratio (ICER) will be calculated as ∆cost/∆effect. QALY will be calculated as life expectancy x HRQoL, as determined by the Danish value set for EQ-5D-5L. Kaplan-Meier estimates will be used for the estimation of median times to clinical recurrence, disease, or death, and their confidence intervals stratified according to follow-up intensity. The difference in clinical recurrence versus molecular recurrence will be compared using paired t-tests and regression analyses.

Data will be analyzed as intention-to-treat and per-protocol. Interim analyses will be made when 50% of patients in each group have been included, and when 100% in each group have been included and have completed a one-year follow-up.

Quality insurance and ethics:

Data completeness and quality will be monitored by the RESPONSE steering committee, and The General Data Protection Regulation, the Danish Data Protection Act, the Health Act, and the Helsinki II declaration will be complied with unconditionally.

The results of the RESPONSE study are expected to be published in international scientific journals. The reporting will follow the CONSORT guidelines for reporting randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated for stage I and low risk stage II colorectal cancer with curative intend.
2. Age 18 years or older.
3. Understands spoken and written Danish language.
4. Able to use digital care-guide as smartphone application.
5. The patient is also included in DANISH.MRD part 1.

Exclusion Criteria:

1. Patients who are unlikely to comply with the protocol, unable to return for subsequent visits and/or otherwise considered by the PIs to be unlikely to complete the study.
2. Patients who are not able or willing to adhere to the digital platform.
3. Patients treated only with local endoscopic resection, e.g.,Transanal Endoscopic microsurgery (TEM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Health related Quality of Life (HRQoL) | At 3 and 5 years follow-up.
  The outcome will be evaluated by EORTC QLQ-C30 - Global. The overall difference between the IG and SG will be calculated, with a score difference of 7 or more considered the minimal clinically important difference (MID).

SECONDARY OUTCOMES:
Overall survival (OS) | At 3 and 5 years follow-up
  Measured as time from surgery to death from any cause. Results from IG will be compared to results from SG.
Recurrence-free survival (RFS) | At 3 and 5 years follow-up.
  Measured as time from surgery until loco-regional recurrence and/or distant metastases, and/or sudden death from colorectal cancer recurrence.
  Time to molecular recurrence will be calculated as the time from no detectable ctDNA until the time of detectable ctDNA. Results from IG will be compared to results from SG.
HRQoL evaluated by EORTC QLQ-C30 for the five functional scales | At 12 and 36 months.
  Evaluation of HRQol will be performed using the EORTC QLQ-C30 for the five functional scales. Differences between IG and SG will be calculated.
HRQoL evaluated by EQ-5D-5L - EUROQOL - 5 Dimensions 5 Levels | At 12 and 36 months.
  Evaluation of HRQol will be performed using the EQ-5D-5L - EUROQOL - 5 Dimensions 5 Levels. Differences between IG and SG will be calculated.
Fear of Cancer Recurrence Inventory score | At 12 and 36 months.
  This will be evaluated by the validated ePROM, FCRI, according to the questionnaire instructions. Results from IG will be compared to results from SG.
ePROM response rates | From 3 to 36 months.
  The response rates and the use of non-digital means and/or support to fulfill questionnaires will be analyzed to evaluate the feasibility of the digital strategy.
Health care cost | At 3 and 5 years.
  The difference in health care cost between IG and SG will be compared to investigate whether the new follow-up program is more costly than standard of care.
Societal costs | At 3 and 5 years.
  The difference in societal cost between IG and SG will be compared.
Quality-adjusted life years (QALYs) | At 3 and 5 years.
  The difference in quality-adjusted life years (QALYs) between IG and SG will be compared.
Patient satisfaction | From 3 to 36 months.
  Patient satisfaction with the follow-up programs will measured by seven validated questions from the national Danish patient satisfaction database, and compared between IG and SG
Prognostic value of ctDNA | At months 3, 12, 24, and 36 after operation
  ctDNA as predictor of CRC recurrence will be evaluated by prospective and retrospective analysis of collected blood samples
FACIT Fatigue - Functional Assessment of Chronic Illness Therapy - Fatigue scale | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Rectal Cancer Pain Score | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Insomnia severity index (ISI) | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
GAD-7 - General Anxiety Disorder-7 | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
PHQ-9 - Patient Health Questionnaire-9 | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
LARS score - Low Anterior Resection Syndrome Score | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Wexner Incontinence Score | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
St. Marks Incontinence Score | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Bristol Stool Chart | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Patient Assessment of Constipation Symptoms | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Colostomy impact score | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
Rectal Cancer Female Sexuality Score (sexually active only) | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
ICIQ - Male/Female Lower Urinary Tract Symptoms | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects
ILEF-5 - International Index for Erectile Function | At 12 and 36 months.
  Used to evaluate organ-specfic and biopsychosocial late effects

OTHER OUTCOMES:
Comparison of cutting edge ctDNA detection methods in plasma. | At 3 and 5 years.
  As new detection methods for ctDNA evolve, we will use plasma from this cohort to comare the techniques side-by-side, to determine which detection method is best suited for commercial use in a Danish setting.

CONTACTS AND LOCATIONS:
Overall Officials: Lene H Iversen, Prof., Principal Investigator — University of Aarhus; Peter Christensen, Prof., Principal Investigator — Aarhus University Hospital; Ole Thorlacius-Ussing, Prof., Principal Investigator — Aalborg University Hospital; Robert Zacchariae, Prof., Principal Investigator — Aarhus University Hospital; Liza Sopina, Ass.Prof., Principal Investigator — University of Southern Denmark; Claus L Andersen, Prof., Principal Investigator — University of Aarhus
Locations (10):
- Denmark (10):
  - Herlev Hospital, Herlev, Capital Region of Denmark
  - Gødstrup Hospital, Herning, Central Jutland
  - Regional Hospital Randers, Randers, Central Jutland
  - Aalborg University Hospital, Aalborg, North Denmark
  - Odense University Hospital, Odense, The Region of Southern Denmark
  - Svendborg Sygehus, Svendborg, The Region of Southern Denmark
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Regional Hospital Horsens, Horsens
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No
Due to Danish law, individual data cannot be shared with other researchers unless it is in a anonymized form. Anonymous data can be shared upon reasonable request to the PIs after the study results have been published.

REFERENCES:
- [Background] DCCG. (DCCG, 2020).
- [Background] DCCG. DCCG'S Nationale retningslinier for diagnostik og behandling af kolorektal cancer - postoperativ kontrol. (2012).
- [Background] Boysen AK, Spindler KL, Hoyer M, Mortensen FV, Christensen TD, Farkas DK, Ording AG. Metastasis directed therapy for liver and lung metastases from colorectal cancer-A population-based study. Int J Cancer. 2018 Dec 15;143(12):3218-3226. doi: 10.1002/ijc.31626. Epub 2018 Oct 22. PMID 29923284
- [Background] Engstrand J, Nilsson H, Stromberg C, Jonas E, Freedman J. Colorectal cancer liver metastases - a population-based study on incidence, management and survival. BMC Cancer. 2018 Jan 15;18(1):78. doi: 10.1186/s12885-017-3925-x. PMID 29334918
- [Background] Franko J, Shi Q, Meyers JP, Maughan TS, Adams RA, Seymour MT, Saltz L, Punt CJA, Koopman M, Tournigand C, Tebbutt NC, Diaz-Rubio E, Souglakos J, Falcone A, Chibaudel B, Heinemann V, Moen J, De Gramont A, Sargent DJ, Grothey A; Analysis and Research in Cancers of the Digestive System (ARCAD) Group. Prognosis of patients with peritoneal metastatic colorectal cancer given systemic therapy: an analysis of individual patient data from prospective randomised trials from the Analysis and Research in Cancers of the Digestive System (ARCAD) database. Lancet Oncol. 2016 Dec;17(12):1709-1719. doi: 10.1016/S1470-2045(16)30500-9. Epub 2016 Oct 12. PMID 27743922
- [Background] Chakedis J, Schmidt CR. Surgical Treatment of Metastatic Colorectal Cancer. Surg Oncol Clin N Am. 2018 Apr;27(2):377-399. doi: 10.1016/j.soc.2017.11.010. Epub 2017 Dec 15. PMID 29496096
- [Background] Hansdotter P, Scherman P, Petersen SH, Mikalonis M, Holmberg E, Rizell M, Naredi P, Syk I. Patterns and resectability of colorectal cancer recurrences: outcome study within the COLOFOL trial. BJS Open. 2021 Jul 6;5(4):zrab067. doi: 10.1093/bjsopen/zrab067. PMID 34308474
- [Background] Osterman E, Glimelius B. Recurrence Risk After Up-to-Date Colon Cancer Staging, Surgery, and Pathology: Analysis of the Entire Swedish Population. Dis Colon Rectum. 2018 Sep;61(9):1016-1025. doi: 10.1097/DCR.0000000000001158. PMID 30086050
- [Background] Nors J, Iversen LH, Erichsen R, Gotschalck KA, Andersen CL. Incidence of Recurrence and Time to Recurrence in Stage I to III Colorectal Cancer: A Nationwide Danish Cohort Study. JAMA Oncol. 2024 Jan 1;10(1):54-62. doi: 10.1001/jamaoncol.2023.5098. PMID 37971197
- [Background] Tarazona N, Gimeno-Valiente F, Gambardella V, Zuniga S, Rentero-Garrido P, Huerta M, Rosello S, Martinez-Ciarpaglini C, Carbonell-Asins JA, Carrasco F, Ferrer-Martinez A, Bruixola G, Fleitas T, Martin J, Tebar-Martinez R, Moro D, Castillo J, Espi A, Roda D, Cervantes A. Targeted next-generation sequencing of circulating-tumor DNA for tracking minimal residual disease in localized colon cancer. Ann Oncol. 2019 Nov 1;30(11):1804-1812. doi: 10.1093/annonc/mdz390. PMID 31562764
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Chen G, Peng J, Xiao Q, Wu HX, Wu X, Wang F, Li L, Ding P, Zhao Q, Li Y, Wang D, Shao Y, Bao H, Pan Z, Ding KF, Cai S, Wang F, Xu RH. Postoperative circulating tumor DNA as markers of recurrence risk in stages II to III colorectal cancer. J Hematol Oncol. 2021 May 17;14(1):80. doi: 10.1186/s13045-021-01089-z. PMID 34001194
- [Background] Henriksen TV, Tarazona N, Frydendahl A, Reinert T, Gimeno-Valiente F, Carbonell-Asins JA, Sharma S, Renner D, Hafez D, Roda D, Huerta M, Rosello S, Madsen AH, Love US, Andersen PV, Thorlacius-Ussing O, Iversen LH, Gotschalck KA, Sethi H, Aleshin A, Cervantes A, Andersen CL. Circulating Tumor DNA in Stage III Colorectal Cancer, beyond Minimal Residual Disease Detection, toward Assessment of Adjuvant Therapy Efficacy and Clinical Behavior of Recurrences. Clin Cancer Res. 2022 Feb 1;28(3):507-517. doi: 10.1158/1078-0432.CCR-21-2404. Epub 2021 Oct 8. PMID 34625408
- [Background] Qaderi SM, van der Heijden JAG, Verhoeven RHA, de Wilt JHW, Custers JAE; PLCRC study group. Trajectories of health-related quality of life and psychological distress in patients with colorectal cancer: A population-based study. Eur J Cancer. 2021 Nov;158:144-155. doi: 10.1016/j.ejca.2021.08.050. Epub 2021 Oct 16. PMID 34666216
- [Background] Sun R, Dai Z, Zhang Y, Lu J, Zhang Y, Xiao Y. The incidence and risk factors of low anterior resection syndrome (LARS) after sphincter-preserving surgery of rectal cancer: a systematic review and meta-analysis. Support Care Cancer. 2021 Dec;29(12):7249-7258. doi: 10.1007/s00520-021-06326-2. Epub 2021 Jul 23. PMID 34296335
- [Background] Sinimaki S, Elfeki H, Kristensen MH, Laurberg S, Emmertsen KJ. Urinary dysfunction after colorectal cancer treatment and its impact on quality of life - a national cross-sectional study in women. Colorectal Dis. 2021 Feb;23(2):384-393. doi: 10.1111/codi.15541. Epub 2021 Feb 8. PMID 33481335
- [Background] Kristensen MH, Elfeki H, Sinimaki S, Laurberg S, Emmertsen KJ. Urinary dysfunction after colorectal cancer treatment and impact on quality of life-a national cross-sectional study in males. Colorectal Dis. 2021 Feb;23(2):394-404. doi: 10.1111/codi.15554. Epub 2021 Feb 17. PMID 33524243
- [Background] Bregendahl S, Emmertsen KJ, Lindegaard JC, Laurberg S. Urinary and sexual dysfunction in women after resection with and without preoperative radiotherapy for rectal cancer: a population-based cross-sectional study. Colorectal Dis. 2015 Jan;17(1):26-37. doi: 10.1111/codi.12758. PMID 25156386
- [Background] Juul T, Brauner AB, Drewes AM, Emmertsen KJ, Krogh K, Laurberg S, Lauritzen MB, Thorlacius-Ussing O, Christensen P; Danish Cancer Society Centre for Research on Survivorship and Late Adverse Effects after Cancer in the Pelvic Organs Study Group. Systematic screening for late sequelae after colorectal cancer-a feasibility study. Colorectal Dis. 2021 Feb;23(2):345-355. doi: 10.1111/codi.15519. Epub 2021 Feb 5. PMID 33420746
- [Background] Tauber NM, Zachariae R, Jensen AB, Thewes B, Skyt I, Elkjaer E, Butow PN, O'Toole MS. ConquerFear-group: Feasibility study with pilot results of a psychological intervention for fear of cancer recurrence delivered in groups. Psychooncology. 2022 Jan;31(1):30-38. doi: 10.1002/pon.5772. Epub 2021 Aug 3. PMID 34289212
- [Background] Tauber NM, O'Toole MS, Dinkel A, Galica J, Humphris G, Lebel S, Maheu C, Ozakinci G, Prins J, Sharpe L, Smith AB, Thewes B, Simard S, Zachariae R. Effect of Psychological Intervention on Fear of Cancer Recurrence: A Systematic Review and Meta-Analysis. J Clin Oncol. 2019 Nov 1;37(31):2899-2915. doi: 10.1200/JCO.19.00572. Epub 2019 Sep 18. PMID 31532725
- [Background] Johannsen M, O'Connor M, O'Toole MS, Jensen AB, Hojris I, Zachariae R. Efficacy of Mindfulness-Based Cognitive Therapy on Late Post-Treatment Pain in Women Treated for Primary Breast Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Oct 1;34(28):3390-9. doi: 10.1200/JCO.2015.65.0770. Epub 2016 Jun 20. PMID 27325850
- [Background] Zachariae R, Amidi A, Damholdt MF, Clausen CDR, Dahlgaard J, Lord H, Thorndike FP, Ritterband LM. Internet-Delivered Cognitive-Behavioral Therapy for Insomnia in Breast Cancer Survivors: A Randomized Controlled Trial. J Natl Cancer Inst. 2018 Aug 1;110(8):880-887. doi: 10.1093/jnci/djx293. PMID 29471478
- [Background] Nissen ER, O'Connor M, Kaldo V, Hojris I, Borre M, Zachariae R, Mehlsen M. Internet-delivered mindfulness-based cognitive therapy for anxiety and depression in cancer survivors: A randomized controlled trial. Psychooncology. 2020 Jan;29(1):68-75. doi: 10.1002/pon.5237. Epub 2019 Nov 1. PMID 31600414
- [Background] Hovdenak Jakobsen I, Vind Thaysen H, Laurberg S, Johansen C, Juul T; FURCA Steering Group. Patient-led follow-up reduces outpatient doctor visits and improves patient satisfaction. One-year analysis of secondary outcomes in the randomised trial Follow-Up after Rectal CAncer (FURCA). Acta Oncol. 2021 Sep;60(9):1130-1139. doi: 10.1080/0284186X.2021.1950924. Epub 2021 Jul 8. PMID 34238100
- [Background] Region Midtjylland, R. Emento: www.emento.dk (2023).